CLINICAL TRIAL: NCT06442397
Title: Feasibility and Acceptability of an Anti-Inflammatory Lifestyle Intervention for Emerging Adult Cancer Survivors
Brief Title: Anti-Inflammatory Lifestyle Intervention for Emerging Adult Cancer Survivors
Acronym: HEAL
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll a sufficient number of participants to launch a cohort despite increased recruitment efforts
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-24-21095; HM20029744 (Other: Virginia Commonwealth University)
Record Dates: First submitted 2024-05-28; First posted 2024-06-04 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Survivorship
Keywords: Adult Cancer Survivors; Anti-Inflammatory Lifestyle for Cancer Survivors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-Inflammatory Lifestyle Intervention (Experimental): A 16-week program consisting of 12 75-minute virtual group meetings
  Interventions: Behavioral: Anti-Inflammatory Lifestyle Intervention

INTERVENTIONS:
Behavioral: Anti-Inflammatory Lifestyle Intervention — Content includes training in empirically-supported strategies to improve psychological function (e.g., restructuring negative thoughts, distress tolerance), with a focus on changing discrete behaviors linked to inflammation (e.g., sleep, processed foods, physical activity), all intertwined with evidence-based behavior change content adapted to meet the needs of EACS. Participants will also receive digital tools to facilitate daily self-monitoring (Fitbit activity monitor, wireless scales, self-monitoring app) and generate information for tailored weekly e-coaching

SUMMARY:
To test the feasibility and acceptability of AILI and associated research procedures among emerging adult cancer survivors (EACS, N=16) age 18-29.

DETAILED DESCRIPTION:
This is a single-arm pilot trial designed to assess the feasibility and acceptability of an anti-inflammatory lifestyle intervention (AILI) for emerging adults (EA) adapted for emerging adult cancer survivors (EACS).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-29
* Cancer diagnosis of any type
* Body fat percentage >16.2% for women; >10.6% for men

Exclusion Criteria:

* Individuals receiving active chemotherapy/radiation or those having completed active chemotherapy/radiation within the past 6 months
* Individuals who are currently pregnant or lactating
* Current involvement in a weight loss program or current use of weight loss medication
* Individuals who report any other uncontrolled medical conditions that may pose a safety issue given the recommendations for the diet and unsupervised physical activity (e.g., uncontrolled hypertension)
* Individuals with rheumatologic and gastrointestinal conditions associated with severe systemic inflammation (e.g., rheumatoid arthritis, systemic lupus erythematosus, Crohn's disease)
* Individuals with medical conditions resulting in known perturbations in the hypothalamic-pituitary-adrenal axis (e.g., endogenous hypercortisolemia [Cushing's syndrome] or adrenal insufficiency)
* Individuals who report a heart condition, chest pain during periods of activity or rest, or loss of consciousness as assessed by the Physical Activity Readiness Questionnaire (PAR-Q)
* Report of lifetime diagnosis of Anorexia Nervosa or Bulimia Nervosa, or any compensatory behaviors (vomiting, laxative abuse) within the previous 3 months
* Hospitalization for depression or other psychiatric disorder within the past 12 months
* Report of lifetime diagnosis of bipolar disorder or psychotic disorder
* Indication of current suicidal intent
* Inability to speak and read English

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10-30 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Test the feasibility of Anti-Inflammatory Lifestyle Intervention (AILI) and associated research procedures among emerging adult cancer survivors (EACS) age 18-29 | Day 0, At end of recruitment period
  The percentage of participants that enroll
Test the feasibility of AILI and associated research procedures among EACS age 18-29 | 4 months
  The percentage of participants that complete the post intervention questionnaire
Test the feasibility of Anti-Inflammatory Lifestyle Intervention (AILI) and associated research procedures among EACS age 18-29. | 4 months
  The percentage of participants that complete the post intervention blood draw
Assess the acceptability of AILI and associated research procedures among EACS age 18-29. | 4 months
  The percentage of participants that complete all study sessions
Assess the acceptability of AILI and associated research procedures among EACS age 18-29. | 4 months
  The percentage of participants that wear the Fitbit >/= 60% throughout the intervention period.
Assess the acceptability of AILI and associated research procedures among EACS age 18-29. | 4 months
  Intervention satisfaction ratings>/= 4 on a 1-5 Likert scale at 4 months, where (1) Strongly Disagree; (2) Disagree; (3) Neither Agree nor Disagree; (4) Agree; (5) Strongly Agree.
Assess the acceptability of AILI and associated research procedures among EACS age 18-29. | 4 months
  Research procedure satisfaction ratings>/= 3 on a 1-5 Likert scale, where (1) Strongly Disagree; (2) Disagree; (3) Neither Agree nor Disagree; (4) Agree; (5) Strongly Agree.

CONTACTS AND LOCATIONS:
Overall Officials: Autumn Lanoye, Ph.D, Principal Investigator — Virginia Commonwealth University

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data at this time.